CLINICAL TRIAL: NCT01996826
Title: A Multi-Center Study of the Safety and Efficacy of Bevacizumab in High-Risk Corneal Transplant Survival
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Reza Dana, MD (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Bascom Palmer Eye Institute (Other); New York Presbyterian Hospital (Other)
Responsible Party: Sponsor-Investigator, Reza Dana, MD, Director, Cornea and Refractive Surgery Service, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-113H
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Corneal Neovascularization; Corneal Graft Failure
Keywords: Corneal Neovascularization; Cornea Blood Vessels; Corneal Graft Failure; High-Risk Penetrating Keratoplasty; Corneal Transplant
MeSH Terms: conditions — Corneal Neovascularization | interventions — Bevacizumab; Carboxymethylcellulose Sodium; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Avastin® (bevacizumab) (Active Comparator): Treatment will begin on Day 0, immediately upon the conclusion of the penetrating keratoplasty procedure with an injection of 0.1 mL (2.5 mg) bevacizumab. Starting Day 1 post-transplant surgery, subjects will begin treatment with topical bevacizumab (1% solution). Topical treatment will be self-administered 4 times a day for 4 weeks.
  The study treatments are to be given in addition to standard of care treatments. Also, all patients will follow a standard post-operative follow-up visit schedule.
  Interventions: Drug: Avastin® (bevacizumab)
- 0.9% NaCl & Refresh Liquigel (Placebo Comparator): Treatment will begin on Day 0, immediately upon the conclusion of the penetrating keratoplasty procedure with an injection of 0.1 mL 0.9% NaCl. Starting Day 1 post-transplant surgery, subjects will begin treatment with topical Refresh Liquigel. Topical treatment will be self-administered 4 times a day for 4 weeks.
  The study treatments (both topical and subconjunctival injection) are to be given in addition to standard of care treatments. Also, all patients will follow a standard post-operative follow-up visit schedule.
  Interventions: Drug: 0.9% NaCl & Refresh Liquigel

INTERVENTIONS:
Drug: Avastin® (bevacizumab) — One time subconjunctival injection of 0.1 mL (2.5 mg) bevacizumab followed by topical treatment with 1% solution bevacizumab four times a day for four weeks.
  Other Names: Avastin®; bevacizumab
  Arms: Avastin® (bevacizumab)
Drug: 0.9% NaCl & Refresh Liquigel — One-time subconjunctival injection of 0.1mL 0.9% NaCl followed by topical treatment with Refresh Liquigel four times a day for four weeks.
  Other Names: Sodium Chloride; Refresh Liquigel; NaCL
  Arms: 0.9% NaCl & Refresh Liquigel

SUMMARY:
The goal of this study is to investigate whether using bevacizumab (Avastin®) is both safe and effective at decreasing the likelihood of a high-risk corneal graft rejection. Patients who are "high-risk" for rejection have blood vessels growing from the white of the eye into the cornea (clear, front region of the eye). The medication is used at the time of surgery and in the weeks following surgery. Participants have a 50/50 chance at receiving the active study medication or a placebo medication.

DETAILED DESCRIPTION:
The purpose of this study is to test the effectiveness of a drug, bevacizumab (Avastin), in preventing blood vessels that often occur after a corneal transplantation which are considered at "high-risk" for rejection. In many cases these blood vessels lead to the graft rejection and eventual failure of the corneal transplant. It is hoped that this treatment will increase the chances of corneal graft survival.

The medication used in this study is called bevacizumab or Avastin (Genentech, Inc). It works by inhibiting the action of a molecule called vascular endothelial growth factor (VEGF). VEGF is a substance molecule that binds to certain cells to stimulate new blood vessel formation. When VEGF is bound to the drug, it cannot stimulate the formation and growth of new blood vessels. Growth of blood vessels into the cornea is a complication which can worsen the prognosis of your corneal transplant and put the transplant at a higher risk for rejection.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Participant willing and able to provide written informed consent
* Willing and able to comply with study assessments for the full duration of the study
* High-risk characteristics for penetrating keratoplasty:

  1. Presence of corneal NV in one or more quadrants (≥ 3 clock hours NV ≥ 2mm from the limbus) OR
  2. Extension of corneal NV to graft-host junction in a previous failed graft
* In generally good stable overall health

Exclusion Criteria:

* History of Stevens-Johnson syndrome or ocular pemphigoid
* Ocular or periocular malignancy
* Non-healing epithelial defect of at least 0.5x0.5 mm in host corneal bed lasting ≥6 weeks preoperatively
* Uncontrolled glaucoma
* Currently on dialysis
* Has received treatment with anti-VEGF agents (intraocular or systemic) within 45 days of study entry
* Concurrent use of systemic anti-VEGF agents
* Change in topical corticosteroid regimen within 14 days of transplantation
* Use of systemic immunosuppressive for indication other than corneal graft rejection
* Pregnancy (positive pregnancy test) or lactating
* Pre-menopausal women not using adequate contraception (Reliable intrauterine devices, hormonal contraception or a spermicide in combination with a barrier method)
* Uncontrolled hypertension defined as systolic blood pressure (BP) ≥150 or diastolic BP ≥90 mmHg
* History of thromboembolic event within 12 months prior to study entry
* Participation in another simultaneous medical investigation or trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Dana, MD, MPH, MSc, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (3):
- United States (3):
  - Bascom Palmer Eye Institute, Miami, Florida
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - New York Presbyterian Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Avastin® (Bevacizumab): Treatment will begin on Day 0, immediately upon the conclusion of the penetrating keratoplasty procedure with an injection of 0.1 mL (2.5 mg) bevacizumab. Starting Day 1 post-transplant surgery, subjects will begin treatment with topical bevacizumab (1% solution). Topical treatment will be self-administered 4 times a day for 4 weeks.
  The study treatments are to be given in addition to standard of care treatments. Also, all patients will follow a standard post-operative follow-up visit schedule.
  Avastin® (bevacizumab): One time subconjunctival injection of 0.1 mL (2.5 mg) bevacizumab followed by topical treatment with 1% solution bevacizumab four times a day for four weeks.
- 0.9% NaCl & Refresh Liquigel: Treatment will begin on Day 0, immediately upon the conclusion of the penetrating keratoplasty procedure with an injection of 0.1 mL 0.9% NaCl. Starting Day 1 post-transplant surgery, subjects will begin treatment with topical Refresh Liquigel. Topical treatment will be self-administered 4 times a day for 4 weeks.
  The study treatments (both topical and subconjunctival injection) are to be given in addition to standard of care treatments. Also, all patients will follow a standard post-operative follow-up visit schedule.
  0.9% NaCl & Refresh Liquigel: One-time subconjunctival injection of 0.1mL 0.9% NaCl followed by topical treatment with Refresh Liquigel four times a day for four weeks.
Period: Overall Study
Arm/Group | Avastin® (Bevacizumab) | 0.9% NaCl & Refresh Liquigel
Started | 39 | 36
Completed | 32 | 33
Not Completed | 7 | 3
Not completed — Lost to Follow-up | 6 | 2
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Avastin® (Bevacizumab) | 0.9% NaCl & Refresh Liquigel | Total
Number analyzed (Participants) | 39 | 36 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 15 | 36
  >=65 years | 18 | 21 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (13.9) | 65.4 (16.0) | 65 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 21 | 19 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 22 | 25 | 47
  More than one race | 4 | 4 | 8
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 38 | 36 | 74

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Rejection Rate
Description: Endothelial rejection rates in patients in the treatment group and the control group were calculated using the Kaplan-Meier survival curve. The Kaplan-Meier/product limit estimator is a non-parametric statistical test used to show the probability of an event occurring at a given time interval. The Kaplan-Meier estimator is used to show what the probability of corneal transplant rejection (and therefore transplant survival) after administration of the active treatment or control.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Avastin® (Bevacizumab) | 0.9% NaCl & Refresh Liquigel
Number analyzed (Participants) | 36 | 36
Participants | 2 | 5
Statistical Analysis 1: Comparison: Avastin® (Bevacizumab) vs 0.9% NaCl & Refresh Liquigel; Endothelial rejection rates in patients in the treatment group and the control group were calculated using the Kaplan-Meier survival curve. The Kaplan-Meier/product limit estimator is a non-parametric statistical test used to show the probability of an event occurring at a given time interval. The Kaplan-Meier estimator is used to show what the probability of corneal transplant rejection (and therefore transplant survival) after administration of the active treatment or control; Test type: Other — Based on prior studies endothelial rejection episodes tend to occur in the range of about 60% of transplants. We used rates ranging from 50 to 70 % to compute the sample size. We specified the probability of a type 1 error equal to 0.05, study power equal to 80%, a follow-up period of 12 months, and 4% loss to follow-up. Calculations resulted in sample size estimates of between 65 and 124 participants; p = 0.10, Log Rank; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.12 to 1.14]

2. Primary Outcome: Number of Participants Experiencing Ocular Adverse Events
Description: Incidence and severity of ocular adverse events during the study (based on ophthalmic examination and subject self-reporting).
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Avastin® (Bevacizumab) | 0.9% NaCl & Refresh Liquigel
Number analyzed (Participants) | 36 | 36
Participants
  Incidence of Ocular Adverse Events | 34 | 35
  Incidence of Mild Ocular Adverse Events | 21 | 21
  Incidence of Moderate Ocular Adverse Events | 8 | 8
  Incidence of Severe Ocular Adverse Events | 4 | 6
Statistical Analysis 1: Comparison: Avastin® (Bevacizumab) vs 0.9% NaCl & Refresh Liquigel; The incidence of Ocular Adverse Events for subjects in intervention group (Avastin® (bevacizumab) and control group (0.9% NaCl & Refresh Liquigel) were counted and compared; Test type: Other — The count of ocular adverse events for subjects in intervention group (Avastin® (bevacizumab) and control group (0.9% NaCl & Refresh Liquigel) were counted and compared; p = 0.36, Fisher Exact; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.78 to 1.06]
Statistical Analysis 2: Comparison: Avastin® (Bevacizumab) vs 0.9% NaCl & Refresh Liquigel; The number of mild severity Ocular Adverse Events for subjects in intervention group (Avastin® (bevacizumab) and control group (0.9% NaCl & Refresh Liquigel) were counted and compared; Test type: Other — Mild ocular adverse events for subjects in intervention group and control group were counted and compared; p = 0.82, Fisher Exact; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.63 to 1.4]
Statistical Analysis 3: Comparison: Avastin® (Bevacizumab) vs 0.9% NaCl & Refresh Liquigel; The number of moderate severity Ocular Adverse Events for subjects in intervention group (Avastin® (bevacizumab) and control group (0.9% NaCl & Refresh Liquigel) were counted and compared; Test type: Other — Moderate severity ocular adverse events for subjects in intervention group and control group were counted and compared; p > 0.99, Fisher Exact; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.41 to 2.2]
Statistical Analysis 4: Comparison: Avastin® (Bevacizumab) vs 0.9% NaCl & Refresh Liquigel; Severe ocular adverse events for subjects in intervention group and control group were counted and compared; Test type: Other — Severe ocular adverse events for subjects in intervention group and control group were counted and compared; p = 0.51, Fisher Exact; Risk Ratio (RR) = 0.63, 95% CI 2-sided [0.20 to 1.9]

3. Primary Outcome: Incidence of Systemic Adverse Events
Description: Incidence and severity of systemic adverse events during the study (based on physical examination, subject self-reporting, and changes in vital sign).
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Avastin® (Bevacizumab) | 0.9% NaCl & Refresh Liquigel
Number analyzed (Participants) | 36 | 36
Participants
  Incidence of Systemic Adverse Events | 34 | 36
  Incidence of Mild Systemic Adverse Events | 10 | 6
  Incidence of Moderate Systemic Adverse Events | 2 | 1
  Incidence of Severe Systemic Adverse Events | 2 | 1
Statistical Analysis 1: Comparison: Avastin® (Bevacizumab) vs 0.9% NaCl & Refresh Liquigel; Test type: Other — The incidence of Systematic Adverse Events for subjects in intervention group (Avastin® (bevacizumab) and control group (0.9% NaCl & Refresh Liquigel) were calculated and compared; p = 0.24, Fisher Exact; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.79 to 1.02]
Statistical Analysis 2: Comparison: Avastin® (Bevacizumab) vs 0.9% NaCl & Refresh Liquigel; The number of mild systemic Adverse Events for subjects in intervention group (Avastin® (bevacizumab) and control group (0.9% NaCl & Refresh Liquigel) were counted and compared; Test type: Other — Mild severity systemic adverse events for subjects in intervention group and control group were counted and compared; p = 0.40, Fisher Exact; Risk Ratio (RR) = 1.62, 95% CI 2-sided [0.68 to 3.9]
Statistical Analysis 3: Comparison: Avastin® (Bevacizumab) vs 0.9% NaCl & Refresh Liquigel; The number of moderate severity systemic Adverse Events for subjects in intervention group (Avastin® (bevacizumab) and control group (0.9% NaCl & Refresh Liquigel) were counted and compared; Test type: Other — Moderate severity systemic adverse events for subjects in intervention group and control group were counted and compared; p > 0.99, Fisher Exact; Risk Ratio (RR) = 1.95, 95% CI 2-sided [0.26 to 14.5]
Statistical Analysis 4: Comparison: Avastin® (Bevacizumab) vs 0.9% NaCl & Refresh Liquigel; The number of severe systemic Adverse Events for subjects in intervention group (Avastin® (bevacizumab) and control group (0.9% NaCl & Refresh Liquigel) were counted and compared; Test type: Other — Severe systemic adverse events for subjects in intervention group and control group were counted and compared; p > 0.99, Fisher Exact; Risk Ratio (RR) = 1.9, 95% CI 2-sided [0.26 to 14.5]

ADVERSE EVENTS:
Time Frame: 12 months
Description: All the subjects once enrolled into study were followed for the duration of the study (12 months) and examined for systematic and ocular adverse events at every study visit. Any adverse events that discovered by the study staff during the study visits were added to the Adverse Events Log. At every visit study subjects were also asked if any Adverse Events occurred in between study visits.
Arm/Group | Avastin® (Bevacizumab) | 0.9% NaCl & Refresh Liquigel
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/36
Serious Adverse Events (participants affected / at risk) | 2/39 | 4/36
Other Adverse Events (participants affected / at risk) | 34/39 | 35/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avastin® (Bevacizumab) (N=39) | 0.9% NaCl & Refresh Liquigel (N=36)
Atrial fibrillation (subject was hospitalized for 3 days) (Cardiac disorders) | 1 (1) | 0 (0)
Urinary Track Infection (subject hospitalized for 3 days) (Renal and urinary disorders) | 1 (1) | 0 (0)
congestive heart failure (subject hospitalized) (Cardiac disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Infections and infestations) | 0 (0) | 1 (1)
a stroke (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avastin® (Bevacizumab) (N=39) | 0.9% NaCl & Refresh Liquigel (N=36)
AC cells in study eye (Eye disorders) | 1 (1) | 1 (1)
AC cells (OS) (Eye disorders) | 0 (0) | 1 (1)
Acanthamoeba infection in study eye (Eye disorders) | 0 (0) | 1 (1)
Acute graft edema (Eye disorders) | 1 (1) | 0 (0)
Allergic reaction to Bacitracin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Allergic reaction to medications prescribed for congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Back Pain (General disorders) | 0 (0) | 1 (1)
Blurred vision (OD) (Eye disorders) | 1 (1) | 1 (2)
Blurry vision (OS) (Eye disorders) | 1 (2) | 3 (5)
Blurry vision (OU) (Eye disorders) | 0 (0) | 1 (1)
Blurry vision in study eye (Eye disorders) | 0 (0) | 2 (2)
Blurry vision (Eye disorders) | 5 (7) | 1 (1)
Broken sutures (2 broken sutures) (Eye disorders) | 1 (1) | 0 (0)
Burning in study eye (Eye disorders) | 0 (0) | 1 (1)
Central epithelial defect in study eye (Eye disorders) | 1 (1) | 0 (0)
Central scotoma in OD (non-study eye) (Eye disorders) | 0 (0) | 1 (1)
Cloudy vision in study eye (Eye disorders) | 1 (1) | 0 (0)
Cloudy vision (Eye disorders) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Corneal edema (OS) (Eye disorders) | 1 (1) | 0 (0)
Corneal infiltrate near the suture (Eye disorders) | 0 (0) | 1 (1)
Corneal Transplant (Eye disorders) | 0 (0) | 1 (1)
Corneal ulcer (Eye disorders) | 1 (1) | 1 (1)
Dark spot in central vision upon awakening each morning (Eye disorders) | 0 (0) | 1 (1)
Darkening of vision (OD) (Eye disorders) | 0 (0) | 1 (1)
Decrease in vision (Eye disorders) | 1 (2) | 1 (1)
Decrease in vision following intravitreal injection of Eylea (Eye disorders) | 0 (0) | 1 (1)
Descement's folds (OS) (Eye disorders) | 0 (0) | 1 (1)
Difficulty seeing (OU) (Eye disorders) | 1 (1) | 0 (0)
Difficulty/pain with walking caused by recent arthritis (General disorders) | 1 (1) | 0 (0)
Dimming of vision (OD) (Eye disorders) | 0 (0) | 1 (1)
Diplopia & glare at night when driving (OS) (Eye disorders) | 0 (0) | 1 (1)
Discomfort with tearing and burning (Eye disorders) | 1 (1) | 0 (0)
Double vision (OU) (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 6 (7) | 3 (3)
Dry eye from allergies in study eye (Eye disorders) | 0 (0) | 1 (1)
Ear wax in the ear causing pain in the ear and face (Ear and labyrinth disorders) | 1 (1) | 0 (0)
High intraocular pressure (Eye disorders) | 4 (4) | 4 (5)
Low intraocular pressure (Eye disorders) | 0 (0) | 1 (1)
Endothelial (Khodadoust) rejection (Eye disorders) | 0 (0) | 1 (1)
Epithelial defect (Eye disorders) | 1 (1) | 3 (4)
Flashes (Eye disorders) | 0 (0) | 2 (3)
Floaters (Eye disorders) | 2 (3) | 4 (4)
Floaters following a clinical laser procedure (Eye disorders) | 0 (0) | 1 (1)
Floater following intravitreal injection of Eylea (Eye disorders) | 0 (0) | 1 (1)
Foreign body sensation (Eye disorders) | 25 (36) | 15 (22)
Graft rejection (Eye disorders) | 1 (1) | 2 (2)
Green discharge in operative eye (Eye disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 1 (1) | 1 (1)
Headaches due to ocular pain (Eye disorders) | 1 (1) | 0 (0)
Herpes keratitis (General disorders) | 1 (1) | 0 (0)
High blood pressure (General disorders) | 4 (7) | 3 (4)
Hospitalization for shortness of breath with logs of edema in legs and fluid in lungs (General disorders) | 0 (0) | 1 (1)
Increase in the frequency of stinging when instilling eye drops (Eye disorders) | 1 (1) | 0 (0)
Infection from scleral lenses in non-study eye (Eye disorders) | 0 (0) | 1 (1)
Irregular heartbeat (Cardiac disorders) | 0 (0) | 1 (1)
Itchy eye (Eye disorders) | 4 (4) | 2 (2)
Left periocular trauma with an electrical cord plug. No injury to the eye. No symptoms. Subject feel (Eye disorders) | 0 (0) | 1 (1)
Eye lid pain (Eye disorders) | 0 (0) | 1 (1)
Light sensitivity in study eye (Eye disorders) | 1 (1) | 0 (0)
Mild irritation in the operative eye following a Lucentis injection (Eye disorders) | 0 (0) | 1 (1)
Mild edema in graft (Eye disorders) | 1 (1) | 0 (0)
Mild ptosis (OD) (Eye disorders) | 0 (0) | 1 (1)
Nausea (General disorders) | 1 (1) | 2 (3)
Obscured vision in study eye (Eye disorders) | 0 (0) | 1 (1)
Ocular pain (Eye disorders) | 18 (23) | 9 (11)
Ocular ache/pain in outer corner of non-study eye (Eye disorders) | 0 (0) | 1 (1)
Ocular pain the night of the surgery (Eye disorders) | 0 (0) | 1 (1)
Ocular redness (Eye disorders) | 0 (0) | 2 (4)
Patient was hospitalized for urinary track infection (General disorders) | 1 (1) | 0 (0)
Patient went to ER for bronchitis (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 14 (25) | 15 (24)
Post-operative ocular pain (Eye disorders) | 1 (1) | 3 (3)
Post-operative mild graft edema (Eye disorders) | 1 (1) | 3 (3)
Post-operative AC cells (Eye disorders) | 2 (2) | 3 (3)
Post-operative stromal edema (Eye disorders) | 3 (3) | 1 (1)
Post-operative mild irritation and soreness (Eye disorders) | 1 (1) | 0 (0)
Post-operative high intraocular pressure (Eye disorders) | 0 (0) | 1 (1)
Post-operative aching/burning in study eye (Eye disorders) | 1 (1) | 1 (1)
Post-operative epithelial defect (Eye disorders) | 0 (0) | 2 (2)
Post-operative tearing (Eye disorders) | 0 (0) | 2 (2)
Post-operative edema (3+) (Eye disorders) | 0 (0) | 1 (1)
Post-operative wound leak at clock hour 4 (Eye disorders) | 0 (0) | 1 (1)
Post-operative acid reflux (Eye disorders) | 0 (0) | 1 (1)
Post-operative diffuse graft edema (Eye disorders) | 0 (0) | 1 (1)
Post-operative increase in mucus in study eye (Eye disorders) | 0 (0) | 1 (1)
Post-operative light sensitivity (OU) (Eye disorders) | 1 (1) | 0 (0)
Post-operative low Intaocular Pressure (Eye disorders) | 1 (1) | 0 (0)
Post-operative iritis (OS) (Eye disorders) | 1 (1) | 0 (0)
Posterior Capsular Opacity (OS) (Eye disorders) | 0 (0) | 1 (1)
Possible rejection (Eye disorders) | 1 (1) | 0 (0)
Punctate epithelial erosions (OS) (Eye disorders) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 1 (1)
Ring of pink around the eye (Eye disorders) | 0 (0) | 1 (1)
Retinal tear following a clinical laser procedure (Eye disorders) | 0 (0) | 1 (1)
Retained lens cortex inferior (OS) (Eye disorders) | 1 (1) | 0 (0)
Recurrent herpes keratitis (General disorders) | 1 (1) | 0 (0)
Severe ocular pain (Eye disorders) | 2 (2) | 1 (1)
Stromal edema (Eye disorders) | 2 (3) | 3 (3)
Stinging upon instillation (Eye disorders) | 1 (1) | 0 (0)
Shortness of breath and swelling in leg (Eye disorders) | 0 (0) | 1 (1)
bruised eye (Eye disorders) | 1 (1) | 0 (0)
increase in back pain (Eye disorders) | 0 (0) | 1 (1)
scraped leg which became infected and resulted in debridement on July 20th. (Eye disorders) | 1 (1) | 0 (0)
graft failure (Eye disorders) | 1 (1) | 0 (0)
eye feeling heavier/tighter than usual (Eye disorders) | 1 (1) | 0 (0)
fever/flu with redness in eye (Eye disorders) | 0 (0) | 1 (1)
new scrape on leg (General disorders) | 1 (1) | 0 (0)
Subject visited podiatrist as toenail was falling off (General disorders) | 1 (1) | 0 (0)
fungal infection in the OD (Eye disorders) | 1 (1) | 0 (0)
"ping or a pluck" sensation (Eye disorders) | 1 (1) | 0 (0)
vision decreased (Eye disorders) | 0 (0) | 1 (1)
flashes of light (Eye disorders) | 0 (0) | 1 (1)
pain behind non-study eye (Eye disorders) | 1 (1) | 0 (0)
blood in stool (Eye disorders) | 0 (0) | 1 (1)
black strips in vision non-study eye (Eye disorders) | 0 (0) | 1 (1)
increase in leg cramps (General disorders) | 1 (1) | 0 (0)
urinary tract infection (General disorders) | 1 (1) | 0 (0)
seasonal allergies (Eye disorders) | 0 (0) | 1 (1)
hand surgery on his right hand (Eye disorders) | 0 (0) | 1 (1)
open blister on leg, which subject attributes to the CHF (Eye disorders) | 0 (0) | 1 (1)
Sub-epithelial infiltrates (Eye disorders) | 0 (0) | 1 (1)
vertigo, light-headedness, and slight nausea (Eye disorders) | 0 (0) | 1 (1)
headache (General disorders) | 1 (1) | 0 (0)
seeing rust colors when looking at lights (Eye disorders) | 0 (0) | 1 (1)
left pupil appears to be smaller than right (Eye disorders) | 1 (1) | 0 (0)
Superior neurocystic edema (OD) (Eye disorders) | 0 (0) | 1 (1)
Tearing (Eye disorders) | 12 (19) | 17 (27)
Tenderness (OS) (Eye disorders) | 0 (0) | 1 (1)
Trichiatic lashes (Eye disorders) | 1 (1) | 2 (2)
Visual disturbances following a clinical laser procedure (Eye disorders) | 0 (0) | 1 (1)
Wound leak (Eye disorders) | 1 (1) | 0 (0)
Vitreous Hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1)
Ocular burning upon instilling ophthalmic medication (Pred Forte and Vigamox) (Eye disorders) | 1 (1) | 0 (0)
Ocular burning upon using eye drops in study eye (Eye disorders) | 0 (0) | 1 (1)
Ocular discomfort (OD) (Eye disorders) | 1 (1) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 1 (1)
Ocular discomfort when closing eyelids tightly (OS) (Eye disorders) | 1 (1) | 0 (0)
Ocular eye irritation (OD) (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT01996826/Prot_SAP_000.pdf